CLINICAL TRIAL: NCT05101694
Title: Study on the Correlation Between Alveolar Macrophage-derived Autophagosomes and the Severity of Lung Injury in ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, professor, Southeast University, China
Other Study IDs: 2021ZDSYLL215-P01
Record Dates: First submitted 2021-09-25; First posted 2021-11-01 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: ARDS
Keywords: macrophage; autophagosome; gene

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — blood and BALF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the process of acute respiratory distress syndrome (ARDS), alveolar macrophages can secrete a large number of autophagosomes to mediate the inflammatory response of ARDS and aggravate the pathological damage of the lungs. At the same time, the meta-transcriptome can detect the expression of all genes without a reference genome. This study intends to explore that Whether the alveoli macrophage-derived autophagosomes are related to the severity and prognosis of ARDS, and try to construct a recognition model to predict the prognosis of ARDS.

DETAILED DESCRIPTION:
Nowadays, acute respiratory distress syndrome (ARDS) is a major clinical problem in the world. Infection and other factors induce immune cells to release inflammatory mediators, and the following uncontrolled inflammatory response is the fundamental reason for the poor prognosis of ARDS. So, it's important to explore the mechanism of ARDS and reduce lung injury.

In the lung tissue, the activation of alveolar macrophages (including alveolar resident macrophages and macrophages recruited in the blood) is an important way that mediates the ARDS inflammatory response. The previous study of the investigator's team proved that alveolar macrophages could not only directly secrete inflammatory mediators, but also mediated the release of inflammatory factors through the secretion of autophagosomes. At the same time, ARDS has been extensively studied in molecular biology, but the prospective exploration of the relationship between the host response and the development mechanism of ARDS is lacking.

The formation of autophagosomes is the marker of autophagy. In the process of ARDS, alveolar macrophages can secrete a large number of autophagosomes to mediate the inflammatory response of ARDS and aggravate the pathological damage of the lungs. At the same time, the meta-transcriptome can detect the expression of all genes without a reference genome, so it has an irreplaceable advantage in exploring the host's response when pathogenic microorganisms invade the body. The investigators speculate that there may be differences in the host response between patients with different types of ARDS.

However, the above results are derived from cell or animal experiments. It hasn't been known whether autophagosomes could be secreted in the alveoli of ARDS patients, and it has not been proven that whether there is a difference in host response between ARDS patients and controls. Therefore, this study intends to explore that Whether the alveoli macrophage-derived autophagosomes are related to the severity and prognosis of ARDS, and try to construct a recognition model to predict the prognosis of ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old
2. Meet ARDS Berlin diagnostic criteria
3. Artificial airway has been established (tracheal intubation, tracheotomy)
4. Sign informed consent
5. Within 7 days of diagnosis of ARDS

Exclusion Criteria:

1. Younger than 18 years old or older than 85 years old
2. Pregnant women, cancer and immune system diseases
3. There are contraindications for bronchoscopy (poor oxygenation/severe heart disease, cardiac insufficiency/abnormal blood clotting, massive hemoptysis/aortic aneurysm risk of rupture, etc.)
4. Patients undergoing other clinical trials
5. Estimated survival time <24h

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ARDS in the Department of Critical Care Medicine, Zhongda Hospital, Southeast University from October 2021 to May 2022
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The link between the proportion of macrophage-derived autophagosomes in alveolar lavage fluid of ARDS patients with the severity of ARDS | at the first day of enrolling the patients
  Getting these data through Flow cytometer and analyzing the link between these data with the severity of ARDS
Autophagosomes in alveolar lavage fluid of ARDS patients with the prognosis of ARDS | at the twenty-eighth day of enrolling the patients
  Getting these data through Flow cytometer and analyzing the link between these data with the prognosis of ARDS

SECONDARY OUTCOMES:
Autophagosomes and macrophage-derived autophagosomes in blood | day 1，day 3 or day 7
  Getting these data through Flow cytometer and analyzing the link between these data with the prognosis of ARDS
extracellular vesicles | day 1，day 3 or day 7
  extracellular vesicles in alveolar lavage fluid and blood through Flow cytometer
Mortality | During hospitalization
  ICU, 28 day and hospital mortality
length of stay | During hospitalization
  ICU and hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, Dr, Study Director — Southeast University
Locations (1):
- Nanjing Zhong-Da Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all the the data and methods can be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data can be available before June 2023 and can be available for all the time
Access Criteria: liulingdoctor@126.com

REFERENCES:
- [Result] Irish Critical Care Trials Group. Acute lung injury and the acute respiratory distress syndrome in Ireland: a prospective audit of epidemiology and management. Crit Care. 2008;12(1):R30. doi: 10.1186/cc6808. Epub 2008 Feb 29. PMID 18312626
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Liu L, Yang Y, Gao Z, Li M, Mu X, Ma X, Li G, Sun W, Wang X, Gu Q, Zheng R, Zhao H, Ao D, Yu W, Wang Y, Chen K, Yan J, Li J, Cai G, Wang Y, Wang H, Kang Y, Slutsky AS, Liu S, Xie J, Qiu H. Practice of diagnosis and management of acute respiratory distress syndrome in mainland China: a cross-sectional study. J Thorac Dis. 2018 Sep;10(9):5394-5404. doi: 10.21037/jtd.2018.08.137. PMID 30416787
- [Result] Sakr Y, Francois B, Sole-Violan J, Kotfis K, Jaschinski U, Estella A, Leone M, Jakob SM, Wittebole X, Fontes LE, de Melo Gurgel M, Midega T, Vincent JL, Ranieri VM; SOAP and ICON Investigators. Temporal changes in the epidemiology, management, and outcome from acute respiratory distress syndrome in European intensive care units: a comparison of two large cohorts. Crit Care. 2021 Feb 25;25(1):87. doi: 10.1186/s13054-020-03455-8. PMID 33632247
- [Result] Pourfathi M, Kadlecek SJ, Chatterjee S, Rizi RR. Metabolic Imaging and Biological Assessment: Platforms to Evaluate Acute Lung Injury and Inflammation. Front Physiol. 2020 Aug 31;11:937. doi: 10.3389/fphys.2020.00937. eCollection 2020. PMID 32982768
- [Result] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Result] Huang X, Xiu H, Zhang S, Zhang G. The Role of Macrophages in the Pathogenesis of ALI/ARDS. Mediators Inflamm. 2018 May 13;2018:1264913. doi: 10.1155/2018/1264913. eCollection 2018. PMID 29950923
- [Result] Dikic I, Elazar Z. Mechanism and medical implications of mammalian autophagy. Nat Rev Mol Cell Biol. 2018 Jun;19(6):349-364. doi: 10.1038/s41580-018-0003-4. PMID 29618831
- [Result] Mizushima N, Levine B. Autophagy in Human Diseases. N Engl J Med. 2020 Oct 15;383(16):1564-1576. doi: 10.1056/NEJMra2022774. No abstract available. PMID 33053285
- [Result] Wang J, Davis S, Zhu M, Miller EA, Ferro-Novick S. Autophagosome formation: Where the secretory and autophagy pathways meet. Autophagy. 2017 May 4;13(5):973-974. doi: 10.1080/15548627.2017.1287657. Epub 2017 Feb 15. PMID 28287860
- [Result] Gonzalez CD, Resnik R, Vaccaro MI. Secretory Autophagy and Its Relevance in Metabolic and Degenerative Disease. Front Endocrinol (Lausanne). 2020 May 5;11:266. doi: 10.3389/fendo.2020.00266. eCollection 2020. PMID 32477265
- [Result] Davis S, Wang J, Ferro-Novick S. Crosstalk between the Secretory and Autophagy Pathways Regulates Autophagosome Formation. Dev Cell. 2017 Apr 10;41(1):23-32. doi: 10.1016/j.devcel.2017.03.015. PMID 28399396
- [Result] Bel S, Pendse M, Wang Y, Li Y, Ruhn KA, Hassell B, Leal T, Winter SE, Xavier RJ, Hooper LV. Paneth cells secrete lysozyme via secretory autophagy during bacterial infection of the intestine. Science. 2017 Sep 8;357(6355):1047-1052. doi: 10.1126/science.aal4677. Epub 2017 Jul 27. PMID 28751470